CLINICAL TRIAL: NCT07085416
Title: Sensor Ankle Brace for Special Operations Rehabilitation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: TAYCO BRACE, INC (Unknown); United States Air Force (U.S. Federal Agency)
Responsible Party: Principal Investigator, Allison Gruber, PhD, Associate Professor of Kinesiology, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 22304; FWR20240183X (Other: Air Force Protocol Number)
Record Dates: First submitted 2025-06-26; First posted 2025-07-25 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Gait; Balance; Biomechanical Data; Postural Control; Locomotion
Keywords: adult; gait; gait analysis; humans; ankle brace; motion capture; sensor validation; wearable electronic devices; wearable sensors; inertial measurement unit; IMU; locomotion; running; walking; landing; stair ascent; stair descent

STUDY DESIGN:
Intervention Model Description: This is a randomized, open-label, single-group interventional study evaluating the measurement feasibility of the TayCo Brace, Inc. sensor-enabled Athletic X ankle brace (sXAB). The primary purpose of this study is to conduct a clinical trial to test a prototype device for feasibility and not health outcomes. To do so, we will compare gait and balance metrics derived from the sXAB to those from gold-standard motion capture and research-grade inertial measurement units (IMUs). Participants may complete one or both protocols. Protocol/cohort 1 includes a balance test and walking at two speeds with and without the sXAB. Protocol/cohort 2 includes a balance test, stair ascent, stair descent, drop landing, walking, and running, all performed under brace and no-brace conditions. The order of bracing conditions will be randomized for each participant, as will the order of tasks and speeds within each condition. The study is not blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Single Group: Brace and No-Brace Conditions (Experimental): This study includes a single group of participants (collected across two cohorts) who complete movement tasks under two within-subject conditions: (1) wearing a sensor-enabled ankle brace ("brace" condition), and (2) without the brace ("no-brace" condition). Each participant serves as their own control. The brace condition order is randomized, and all participants experience both conditions.
  Interventions: Device: Sensor-enabled Athletic X Ankle Brace (sXAB)

INTERVENTIONS:
Device: Sensor-enabled Athletic X Ankle Brace (sXAB) — The intervention is a sensor-enabled version of the TayCo Brace, Inc. Athletic X Ankle Brace (sXAB), which integrates commercially available inertial measurement units (IMUs) into the structure of the brace. The brace is worn on the ankle of the dominant limb during functional movement tasks to evaluate its ability to produce valid gait and balance metrics compared to laboratory-grade measurement systems.

SUMMARY:
The primary purpose of this study is to conduct a clinical trial to test a prototype device for feasibility and not health outcomes. To do this, the investigators will evaluate the performance of commercially available inertial measurement unit sensors incorporated into an existing ankle brace ("sXAB") by TayCo Brace, Inc. We will compare the gait metrics calculated from the sensors incorporated into the brace with gold-standard equipment that is used in research and clinical settings to determine whether the sXAB performs adequately in terms of measurement or technical feasibility prior to further clinical evaluation. The sensors in the ankle brace will be validated in the lab, first on healthy subjects walking in standard tennis shoes/sneakers (protocol 1), and secondarily in the lab on healthy subjects wearing combat boots performing walking, running, jumping, and stair climbing (protocol 2). These movements were selected because they simulate key movements performed during operational activities. Protocol 1 will take place first, then aspects of the sXAB will be evaluated and implemented, then protocol 2 will take place. Participants completing protocol 1 are eligible to complete protocol 2. The study includes two cohorts of participants completing different functional tasks. All participants experience both conditions: with an ankle brace and without an ankle brace. Comparisons are made within-subject between brace and no-brace conditions. It is hypothesized that the sensor-enabled ankle brace will measure gait metrics with a high degree of accuracy (within 5%) when compared against the gold-standard lab equipment (i.e., motion capture and research-grade inertial measurement units).

DETAILED DESCRIPTION:
This study is funded by a grant from the United States Air Force awarded to TayCo Brace, Inc. The required research partner, Indiana University (Principal Investigator Allison Gruber, PhD), holds the subaward. All human subjects activities are taking place at the Indiana University Bloomington (IUB) campus. Potential participants for study protocols 1 and 2 will be recruited from the community and the IUB campus. Paper flyers will be posted on campus and the surrounding commercial areas. Electronic flyers will be posted in the IUB classifies, on the iConnect website, and on social media. Potential participants will either contact the research team to complete the initial screening or respond to the flyer via a QR code that takes them directly to the online version of the screening form. The screening form asks yes/no questions from the Physical Activity Readiness Questionnaire (PARQ+) and additional questions about the individuals health history, musculoskeletal injury history, and current physical activity levels. After initial screening to determine eligibility, provisionally eligible participants will come to the laboratory on the IUB campus to complete enrollment and study procedures.

During visit 1 for study protocols 1 and 2, participants will read the informed consent document and, after all questions have been answered, sign the informed consent document if they agree to participate in the study. Next, participants will complete a health history questionnaire which repeats the PARQ+ questions and additional health history questions presented in the initial screening to confirm eligibility. Foot length measurements and additional surveys (i.e., the Identification of Functional Ankle Instability (IDFAI) and International Physical Activity Questionnaire - Short Form (IPAQ)) will be administered to confirm eligibility in protocol 2 but for protocol 1 the IDFAI and IPAQ will be collected for informative purposes and to help explain variability between participants. If eligibility is confirmed, participants will be enrolled and complete the study procedures. After eligibility is confirmed, all participants for both protocols will also complete the past-year physical activity questionnaire (PYPAQ) and protocol 2 participants will complete a running history questionnaire.

Following the surveys, height and weight will be measured then the dominant limb test and the preferred speed test will be performed. The dominant limb test determines whether the right or left lower limb is the dominant limb by observing which limb participants use to kick a ball. The preferred speed test involves the participant walking or running at or near their reported preferred speed (or 2.9 mph for walking and 4.5 mph for running if preferred speed is unknown). The speed will be blinded to the participant. The researcher will increase or decrease the speed in 0.5-1.0 mph increments until the participant identifies the same speed as their preferred speed three times.

Next, the participant will be prepared for data collection. Participants will be asked to change into form fitting clothing (provided by the laboratory, if needed) and the shoes they prefer to wear during exercise or physical activity (protocol 1), or combat boots provided by the laboratory (protocol 2). Next, reflective markers and the lab's research-grade inertial measurement units (IMUs) will be placed on anatomical landmarks of both feet, lower-legs, thighs, and pelvis, and the sensor-enabled ankle brace ("sXAB") will be secured on the dominant limb, if the first randomized condition is the brace condition. Participants will warm-up by walking on a treadmill before completing each of the brace conditions (brace and no-brace) to acclimate wearing the brace and/or the reflective markers and lab IMUs. Participants will then be asked to complete the movement tests specific to each protocol (protocol 1: standing balance, walking at preferred speed, walking at a standardized speed of 2.9 mph; protocol 2: standing balance, stairs, drop landing, walking at preferred speed, and running at preferred speed) while wearing the sXAB and without wearing the brace ("no brace" condition) as three-dimensional motion capture data, force plate data, IMU data, and data from the sXAB (if worn) are recorded. The order of the bracing conditions will be presented in a random order. The brace will be worn on the dominant limb. Within each brace condition, the standing balance test will be performed first then the remaining movements will be presented in a random order. After the first brace condition is complete, the participant will be prepared to complete the second brace condition then repeat the warm-up, standing balance test, and the movement tests.

Protocol 1 is expected to begin in late June 2025 and involve N=20 participants. After protocol 1 is complete, TayCo Brace, Inc. will make adjustments to the sXAB such as device placement on the brace, algorithms to output outcome measures, etc. that will be tested during protocol 2. Protocol 2 is expected to begin in September 2025 and will involve N=40 participants. Although device feasibility studies typically involve smaller sample sizes, this study includes a larger cohort (N = 60) to enable evaluation of sensor-derived metrics across a broad range of functional tasks. The study aims to determine whether gait and balance measures obtained from an ankle brace integrated with inertial measurement units are comparable to those from gold-standard laboratory tools, such as motion capture and research-grade IMUs.

The ankle brace used in this study is an FDA Class I exempt device. The version used includes integrated commercially available inertial sensors in which the investigators are evaluating their use with the brace against standard laboratory-based systems. The study does not involve a new intended use or clinical treatment evaluation.

ELIGIBILITY:
Inclusion Criteria for both cohorts:

* Healthy adults: ages 18 - 40 years
* considered "healthy to exercise" as determined by the physical activity readiness questionnaire (PAR-Q)

Additional Inclusion Criteria specific to cohort 2 only:

* Classified as "moderate" or "high" activity level as defined by the scoring criteria of the International Physical Activity Questionnaire - Short Form (IPAQ)
* Comfortably fit into combat boots provided by the laboratory (Men's sizes 8, 9, 10, 11, 12 and Women's sizes 6, 7, 8, 9, 10 will be purchased, and so participants with foot lengths of 22.54-29.27.8 cm are expected to fit in the boots provided).

Exclusion Criteria for both cohorts:

* Smoking tobacco on a regular basis
* Previous lower back or lower limb surgery (including the joints of the pelvis and lower limbs)
* Musculoskeletal injury sustained within the 12-weeks prior to enrollment . A musculoskeletal injury is defined as musculoskeletal pain causing a reduction or stoppage of normal physical activity for at least 3 days within a 7-day period, and have not returned to their normal physical activity and exercise without pain for at least the last 6-weeks.
* Pregnant (women only)
* Current or history of an unresolved musculoskeletal, neurological, cardiovascular, pulmonary/respiratory, metabolic, renal condition, disease, or problem.
* Torn anterior or posterior cruciate ligament (ACL or PCL).
* Any other disease or problems that may affect movement or the ability to exercise even at a low intensity.

Additional Exclusion Criteria specific to cohort 2 only:

* Identification of Functional Ankle Instability (IDFAI) score of <11.
* unable to comfortably perform the drop landing condition.
* Feet are too large or too small to fit comfortably in the combat boots provided.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-16 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-06-18 (Estimated)

PRIMARY OUTCOMES:
Feasibility of collecting valid kinematic data with the sensor-enabled ankle brace (sXAB). | At study visit(s), completed up to 1 week after enrollment.
  This outcome evaluates whether kinematic data collected using the sensor-enabled ankle brace (sXAB) are sufficiently accurate and reliable compared to gold-standard laboratory systems (motion capture, force plates, and research-grade IMUs), thereby supporting feasibility of using the sXAB for measuring these variables. Agreement will be assessed using equivalence testing across variables (e.g., joint angles, range of motion), which will be aggregated into a single equivalence score for kinematics by taking the average and standard deviation across variables. Data are collected during brace and no-brace conditions across multiple movement tasks. Feasibility is supported if equivalence criteria are met for all core variables.
Feasibility of collecting valid spatiotemporal parameters with the sensor-enabled ankle brace (sXAB). | At study visit(s), completed up to 1 week after enrollment.
  This outcome evaluates whether spatiotemporal parameters collected using the sensor-enabled ankle brace (sXAB) are sufficiently accurate and reliable compared to gold-standard laboratory systems (motion capture, force plates, and research-grade IMUs), thereby supporting feasibility of using the sXAB for measuring these variables. Agreement will be assessed using equivalence testing across variables (e.g., stance time, stride length, gait speed), which will be aggregated into a single equivalence score for spatiotemporal parameters by taking the average and standard deviation across variables. Data are collected during brace and no-brace conditions across multiple movement tasks. Feasibility is supported if equivalence criteria are met for all core variables.
Feasibility of collecting valid postural balance data with the sensor-enabled ankle brace (sXAB). | At study visit(s), completed up to 1 week after enrollment.
  This outcome evaluates whether postural balance data collected using the sensor-enabled ankle brace (sXAB) are sufficiently accurate and reliable compared to gold-standard laboratory systems (motion capture, force plates, and research-grade IMUs), thereby supporting feasibility of using the sXAB for measuring these variables. Agreement will be assessed using equivalence testing across variables (e.g., sway amplitude and velocity), which will be aggregated into a single equivalence score for postural balance by taking the average and standard deviation across variables. Data are collected during brace and no-brace conditions across multiple movement tasks. Feasibility is supported if equivalence criteria are met for all core variables.

SECONDARY OUTCOMES:
Feasibility of collecting valid kinetic data with the sensor-enabled ankle brace (sXAB). | At study visit(s), completed up to 1 week after enrollment.
  This outcome evaluates whether kinetic data collected using the sensor-enabled ankle brace (sXAB) are sufficiently accurate and reliable compared to gold-standard laboratory systems (motion capture, force plates, and research-grade IMUs), thereby supporting feasibility of using the sXAB for measuring these variables. Agreement will be assessed using equivalence testing across variables (e.g., peak vertical ground reaction force, total vertical impulse), which will be aggregated into a single equivalence score for kinetics by taking the average and standard deviation across variables. Data are collected during brace and no-brace conditions across multiple movement tasks. Feasibility is supported if equivalence criteria are met for all core variables.
Feasibility of collecting valid wear time with the sensor-enabled ankle brace (sXAB). | At study visit(s), completed up to 1 week after enrollment.
  This outcome evaluates whether wear time collected using the sensor-enabled ankle brace (sXAB) are sufficiently accurate and reliable compared to gold-standard laboratory systems (motion capture, force plates, and research-grade IMUs), thereby supporting feasibility of using the sXAB for measuring these variables. Agreement will be assessed using equivalence testing across variables (e.g., time on and off, total daily wear duration), which will be aggregated into a single equivalence score for wear time by taking the average and standard deviation across variables. Data are collected during brace and no-brace conditions across multiple movement tasks. Feasibility is supported if equivalence criteria are met for all core variables.
Feasibility of valid activity recognition with the sensor-enabled ankle brace (sXAB). | At study visit(s), completed up to 1 week after enrollment.
  This outcome evaluates whether activity recognition assessed from data collected by the sensor-enabled ankle brace (sXAB) are sufficiently accurate and reliable compared to gold-standard laboratory systems (motion capture, force plates, and research-grade IMUs), thereby supporting feasibility of using the sXAB for measuring these variables. Agreement will be assessed using equivalence testing across variables (e.g., start, stop, and total time walking and running), which will be aggregated into a single equivalence score for activity recognition by taking the average and standard deviation across variables. Data are collected during brace and no-brace conditions across multiple movement tasks. Feasibility is supported if equivalence criteria are met for all core variables.

CONTACTS AND LOCATIONS:
Overall Officials: Allison H Gruber, PhD, Principal Investigator — Indiana University
Locations (1):
- Indiana University, School of Public Health - Bloomington, Bloomington, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
The principal investigator will share data summaries and statistical outcomes with TayCo Brace, Inc. to inform improvements to the sXAB device between protocol phases and guide future development. Only de-identified, processed data will be shared. Shared data may include participant demographics (e.g., age, sex, height), survey responses, and data from motion capture, force plates, IMUs, and the sXAB. The U.S. Department of Defense personnel responsible for human subject protections may request access to de-identified research records, which will be provided in their preferred format and method. Data collected in this study may also be used for future research and scholarly publications. All shared or reused data will be de-identified.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: De-identified data will be provided to TayCo Brace, Inc. after completion of each protocol phase (i.e., following Protocol 1 and again after Protocol 2). TayCo Brace, Inc. may retain these data indefinitely for product development purposes. No individual participant data will be publicly posted or shared beyond the research sponsor and authorized personnel.
Access Criteria: Access to individual participant data is limited to authorized personnel at TayCo Brace, Inc. and U.S. Department of Defense research oversight officials. No public access to individual-level data is planned. All data shared will be de-identified and used solely for device development or regulatory oversight purposes. Access to de-identified data for additional research may be considered upon request, subject to institutional approval and data use agreements.

REFERENCES:
- [Background] Rhon DI, Greenlee TA, Cook CE, Westrick RB, Umlauf JA, Fraser JJ. Fractures and Chronic Recurrence are Commonly Associated with Ankle Sprains: a 5-year Population-level Cohort of Patients Seen in the U.S. Military Health System. Int J Sports Phys Ther. 2021 Oct 1;16(5):1313-1322. doi: 10.26603/001c.27912. eCollection 2021. PMID 34631252
- [Background] Gurchiek RD, Choquette RH, Beynnon BD, Slauterbeck JR, Tourville TW, Toth MJ, McGinnis RS. Open-Source Remote Gait Analysis: A Post-Surgery Patient Monitoring Application. Sci Rep. 2019 Nov 29;9(1):17966. doi: 10.1038/s41598-019-54399-1. PMID 31784691
- [Background] Hafer JF, Provenzano SG, Kern KL, Agresta CE, Grant JA, Zernicke RF. Measuring markers of aging and knee osteoarthritis gait using inertial measurement units. J Biomech. 2020 Jan 23;99:109567. doi: 10.1016/j.jbiomech.2019.109567. Epub 2019 Dec 27. PMID 31916999